CLINICAL TRIAL: NCT01399788
Title: An Open Label, Single Dose, 2-Way Cross-Over Randomized Bioequivalence Study Comparing a Fixed Dose Combination Formulation, Myrin®-p Forte, (Contains 150 Mg Rifampicin, 75 Mg Isoniazid, 275 Mg Ethambutol and 400 Mg Pyrazinamide Per Tablet) to an Equivalent Dose of Single Drug Reference Preparations of Rifampicin, Isoniazid, Ethambutol and Pyrazinamide Following Oral Administration in Healthy Adults Under Fasting Conditions
Brief Title: A Bioequivalence Study Comparing A Fixed Dose Combination Formulation Of Myrin P Forte That Contains Rifampicin, Isoniazid, Ethambutol And Pyrazinamide Per Tablet To An Equivalent Dose Of Single Drug Reference Preparations Of Similar Combination Following Oral Administration In Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: B3801002
Record Dates: First submitted 2011-07-13; First posted 2011-07-22 (Estimated); Results first posted 2012-03-16 (Estimated); Last update posted 2017-04-05 (Actual); Status verified 2017-03

CONDITIONS: Healthy Volunteers
Keywords: Bioequivalence; Healthy Volunteers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1.0 (Active Comparator): Test Myrin P Forte Contains 150mg Rifampicin, 75mg Isoniazid, 275mg Ethambutol, 400mg Pyrazinamide
  Interventions: Drug: Myrin P Forte
- 2.0 (Active Comparator): Reference Single drug reference preparations contain Rifampicin, Isoniazid, Ethambutol, Pyrazinamide
  Interventions: Drug: Single drug references

INTERVENTIONS:
Drug: Myrin P Forte — Tablet containing Rifampicin, Isoniazid, Ethambutol and Pyrazinamide, given once daily, single dose
  Arms: 1.0
Drug: Single drug references — containing Rifampicin, Isoniazid, Ethambutol and Pyrazinamide as single agents
  Arms: 2.0

SUMMARY:
This is a bioequivalence trial to evaluate the bioequivalence of Myrin P Forte against reference drug in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, male or female, 21 to 55 years of age, body weight no less than 55 kg, Body mass index (BMI) of 17.5 to 30.5 kg/m2. Healthy is defined as no clinically relevant abnormalities identified by a detailed medical history, full physical examination, including blood pressure and pulse rate measurement, 12-lead electrocardiogram (ECG) or clinical laboratory tests.
* An informed consent document signed and dated by the subject.
* Subjects who are willing and able to comply with all scheduled visits, treatment plan, laboratory tests, and other study procedures.

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at the time of dosing), positive Hepatitis B surface antigen or Human Immunodeficiency Virus (HIV) serology results.
* pregnant or nursing female,
* alcohol, drug, smoke user,
* sensitive to any study medication or related component,
* History or active gout,
* History or active tuberculosis,
* Known optic neuritis or other ophthalmological conditions.

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2011-07; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Singapore, Singapore

REFERENCES:
- [Derived] Wang HF, Wang R, O'Gorman M, Crownover P, Naqvi A, Jafri I. Bioequivalence of fixed-dose combination Myrin(R)-P Forte and reference drugs in loose combination. Int J Tuberc Lung Dis. 2013 Dec;17(12):1596-601. doi: 10.5588/ijtld.13.0190. PMID 24200275

RESULTS

PARTICIPANT FLOW:
Groups:
- Myrin-P Forte First, Then Four Single Drug References: Single oral dose of 4 fixed dose combination (FDC) tablets of Myrin-P Forte (each tablet contains 150 milligram (mg) rifampicin, 75 mg isoniazid, 275 mg ethambutol and 400 mg pyrazinamide) in first intervention period; and single oral dose of 4 reference products: 600 mg rifampicin capsules, 300 mg isoniazid, 1100 mg ethambutol and 1500 mg pyrazinamide tablets in second intervention period. A washout period of at least 1 week was maintained between each period.
- Four Single Drug References First, Then Myrin-P Forte: Single oral dose of 4 reference products: 600 mg rifampicin capsules, 300 mg isoniazid, 1100 mg ethambutol and 1500 mg pyrazinamide tablets in first intervention period; and single oral dose of 4 FDC tablets of Myrin-P Forte (each tablet contains 150 mg rifampicin, 75 mg isoniazid, 275 mg ethambutol and 400 mg pyrazinamide) in second intervention period. A washout period of at least 1 week was maintained between each period.
Period: First Intervention Period
Arm/Group | Myrin-P Forte First, Then Four Single Drug References | Four Single Drug References First, Then Myrin-P Forte
Started | 18 | 18
Completed | 17 | 18
Not Completed | 1 | 0
Not completed — Adverse Event | 1 | 0
Period: Washout Period (at Least 1 Week)
Arm/Group | Myrin-P Forte First, Then Four Single Drug References | Four Single Drug References First, Then Myrin-P Forte
Started | 17 | 18
Completed | 17 | 18
Not Completed | 0 | 0
Period: Second Intervention Period
Arm/Group | Myrin-P Forte First, Then Four Single Drug References | Four Single Drug References First, Then Myrin-P Forte
Started | 17 | 18
Completed | 17 | 18
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Entire Study Population: Includes participants randomized to receive Myrin-P Forte first and four single drug references first.
Arm/Group | Entire Study Population
Number analyzed (Participants) | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.6 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 34

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast)
Description: Area under the plasma concentration-time curve from time zero (pre-dose) to the time of last measured concentration (AUClast).
Time Frame: 0 (pre-dose), 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 16 and 24 hours (hrs) post-dose
Population: Pharmacokinetic (PK) parameter analysis population included all randomized and treated participants who had at least 1 of the PK parameters for one of four analytes in at least 1 treatment period.
Measure: Geometric Mean (Standard Deviation); unit: ng*hr/mL
Groups:
- Myrin-P Forte: Single oral dose of 4 FDC tablets of Myrin-P Forte (Test) in either first intervention period or second intervention period. Each tablet contains 150 mg rifampicin, 75 mg isoniazid, 275 mg ethambutol and 400 mg pyrazinamide.
- Four Single Drug References: Single oral dose of 4 reference products: 600 mg rifampicin capsules, 300 mg isoniazid, 1100 mg ethambutol and 1500 mg pyrazinamide tablets in either first intervention period or second intervention period.
Arm/Group | Myrin-P Forte | Four Single Drug References
Number analyzed (Participants) | 36 | 35
ng*hr/mL
  Rifampicin | 79360.0 (29613.0) | 77180.0 (20516.0)
  Isoniazid | 20550.0 (12920.0) | 18800.0 (12941.0)
  Ethambutol | 15070.0 (3298.8) | 15170.0 (3119.1)
Statistical Analysis 1: Comparison: Myrin-P Forte vs Four Single Drug References; Rifampicin; 32 participants (16 per sequence) provided at least 99% power that 90% confidence interval (CI) for ratio of test to reference for AUClast lie within acceptance region of 80% - 125%. An intra-subject coefficient of variation (CV) estimate of approximately 14.5% for AUClast was used for this power calculation. Natural log transformed AUClast was analyzed using mixed effect model with sequence, period and treatment as fixed effects and participant within sequence as a random effect; Test type: Superiority or Other; Ratio of Adjusted Means = 103.81, 90% CI 2-sided [99.20 to 108.64]
Statistical Analysis 2: Comparison: Myrin-P Forte vs Four Single Drug References; Isoniazid; 32 participants (16 per sequence) provided at least 99% power that 90% CI for ratio of test to reference for AUClast lie within acceptance region of 80% - 125%. An intra-subject CV estimate of approximately 12.0% for AUClast was used for this power calculation. Natural log transformed AUClast was analyzed using mixed effect model with sequence, period and treatment as fixed effects and participant within sequence as a random effect; Test type: Superiority or Other; Ratio of Adjusted Means = 107.28, 90% CI 2-sided [101.95 to 112.90]
Statistical Analysis 3: Comparison: Myrin-P Forte vs Four Single Drug References; Ethambutol; 32 participants (16 per sequence) provided at least 99% power that 90% CI for ratio of test to reference for AUClast lie within acceptance region of 80% - 125%. An intra-subject CV estimate of approximately 12.9% for AUClast was used for this power calculation. Natural log transformed AUClast was analyzed using mixed effect model with sequence, period and treatment as fixed effects and participant within sequence as a random effect; Test type: Superiority or Other; Ratio of Adjusted Means = 99.48, 90% CI 2-sided [94.92 to 104.25]

2. Primary Outcome: Maximum Observed Plasma Concentration (Cmax)
Time Frame: 0 (pre-dose), 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 16 and 24 hrs post-dose
Population: PK parameter analysis population included all randomized and treated participants who had at least 1 of the PK parameters for one of four analytes in at least 1 treatment period.
Measure: Geometric Mean (Standard Deviation); unit: ng/mL
Arm/Group | Myrin-P Forte | Four Single Drug References
Number analyzed (Participants) | 36 | 35
ng/mL
  Rifampicin | 12120.0 (3682.3) | 11830.0 (2351.8)
  Isoniazid | 4418.0 (1619.0) | 4237.0 (1658.9)
  Ethambutol | 2771.0 (825.4) | 2865.0 (950.5)
Statistical Analysis 1: Comparison: Myrin-P Forte vs Four Single Drug References; Rifampicin: 32 participants (16 per sequence) provided at least 98% power that 90% CI for ratio of test to reference for Cmax lie within acceptance region of 80% - 125%. An intra-subject CV estimate of approximately 18.2% for Cmax was used for this power calculation. Natural log transformed Cmax was analyzed using mixed effect model with sequence, period and treatment as fixed effects and participant within sequence as a random effect; Test type: Superiority or Other; Ratio of Adjusted Means = 102.75, 90% CI 2-sided [95.36 to 110.71]
Statistical Analysis 2: Comparison: Myrin-P Forte vs Four Single Drug References; Isoniazid; 32 participants (16 per sequence) provided at least 98% power that 90% CI for ratio of test to reference for Cmax lie within acceptance region of 80% - 125%. An intra-subject CV estimate of approximately 18.2% for Cmax was used for this power calculation. Natural log transformed Cmax was analyzed using mixed effect model with sequence, period and treatment as fixed effects and participant within sequence as a random effect; Test type: Superiority or Other; Ratio of Adjusted Means = 103.85, 90% CI 2-sided [92.13 to 117.07]
Statistical Analysis 3: Comparison: Myrin-P Forte vs Four Single Drug References; Ethambutol; 32 participants (16 per sequence) provided at least 99% power that 90% CI for ratio of test to reference for Cmax lie within acceptance region of 80% - 125%. An intra-subject CV estimate of approximately 16.0% for Cmax was used for this power calculation. Natural log transformed Cmax was analyzed using mixed effect model with sequence, period and treatment as fixed effects and participant within sequence as a random effect; Test type: Superiority or Other; Ratio of Adjusted Means = 99.48, 90% CI 2-sided [94.92 to 104.25]

3. Primary Outcome: Dose Normalized Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast[dn]) for Pyrazinamide
Description: AUClast[dn] = Dose normalized area under the plasma concentration-time curve (AUC[dn]) from time zero (pre-dose) to the time of last measured concentration. It is obtained from AUClast divided by dose and then multiplied by 1500. The test and reference for pyrazinamide were given at different doses, so dose-normalized parameters were used for analysis for adjusting the dose effect on bioequivalence conclusion.
Time Frame: 0 (pre-dose), 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 16, 24, 36 and 48 hrs post-dose
Population: as for outcome 2
Measure: Geometric Mean (Standard Deviation); unit: (ng*hr/mL)/mg
Arm/Group | Myrin-P Forte | Four Single Drug References
Number analyzed (Participants) | 36 | 35
(ng*hr/mL)/mg | 453500 (76250) | 447900 (82578)
Statistical Analysis 1: Comparison: Myrin-P Forte vs Four Single Drug References; Pyrazinamide; 32 participants (16 per sequence) provided at least 99% power that 90% CI for ratio of test to reference for AUClast lie within acceptance region of 80% - 125%. An intra-subject CV estimate of approximately 5.2% for AUClast was used for this power calculation. Natural log transformed AUClast(dn) was analyzed using mixed effect model with sequence, period and treatment as fixed effects and participant within sequence as a random effect; Test type: Superiority or Other; Ratio of Adjusted Means = 101.73, 90% CI 2-sided [99.12 to 104.40]

4. Primary Outcome: Dose Normalized Maximum Observed Plasma Concentration (Cmax[dn]) for Pyrazinamide
Description: It is obtained from Cmax divided by dose and then multiplied by 1500. The test and reference for pyrazinamide were given at different doses, so dose-normalized parameters were used for analysis for adjusting the dose effect on bioequivalence conclusion.
Time Frame: 0 (pre-dose), 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 16, 24, 36 and 48 hrs post-dose
Population: as for outcome 2
Measure: Geometric Mean (Standard Deviation); unit: (ng/mL)/mg
Arm/Group | Myrin-P Forte | Four Single Drug References
Number analyzed (Participants) | 36 | 35
(ng/mL)/mg | 33890.0 (6490.2) | 35580.0 (12134.0)
Statistical Analysis 1: Comparison: Myrin-P Forte vs Four Single Drug References; Pyrazinamide; 32 participants (16 per sequence) provided at least 99% power that 90% CI for ratio of test to reference for Cmax lie within acceptance region of 80% - 125%. An intra-subject CV estimate of approximately 6.7% for Cmax was used for this power calculation. Natural log transformed Cmax(dn) was analyzed using mixed effect model with sequence, period and treatment as fixed effects and participant within sequence as a random effect; Test type: Superiority or Other; Ratio of Adjusted Means = 95.17, 90% CI 2-sided [88.60 to 102.22]

5. Secondary Outcome: Area Under the Curve From Time Zero to Extrapolated Infinite Time (AUC[0-∞])
Description: AUC (0-∞) = Area under the plasma concentration versus time curve (AUC) from time zero (pre-dose) to extrapolated infinite time (0-∞). It is obtained from AUC (0-t) plus AUC (t-∞).
Time Frame: 0 (pre-dose), 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 16 and 24 hrs post-dose
Population: PK parameter analysis population included all randomized and treated participants who had at least 1 of the PK parameters for one of four analytes in at least 1 treatment period. Here, 'n' is number of participants who were evaluable for this measure.
Measure: Geometric Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Myrin-P Forte | Four Single Drug References
Number analyzed (Participants) | 36 | 35
ng*hr/mL
  Rifampicin (n= 36, 35) | 80940.0 (34613.0) | 78400.0 (22226.0)
  Isoniazid (n= 35, 35) | 21210.0 (13562.0) | 19460.0 (14171.0)
  Ethambutol (n= 28, 31) | 17150.0 (3362.1) | 17050.0 (3378.9)
Statistical Analysis 1: Comparison: Myrin-P Forte vs Four Single Drug References; Rifampicin; Natural log transformed AUC(0-∞) was analyzed using a mixed effect model with sequence, period and treatment as fixed effects and participant within sequence as a random effect; Test type: Superiority or Other; Ratio of Adjusted Means = 104.30, 90% CI 2-sided [99.70 to 109.10]
Statistical Analysis 2: Comparison: Myrin-P Forte vs Four Single Drug References; Isoniazid; Natural log transformed AUC(0-∞) was analyzed using a mixed effect model with sequence, period and treatment as fixed effects and participant within sequence as a random effect; Test type: Superiority or Other; Ratio of Adjusted Means = 105.74, 90% CI 2-sided [100.32 to 111.46]
Statistical Analysis 3: Comparison: Myrin-P Forte vs Four Single Drug References; Ethambutol; Natural log transformed AUC(0-∞) was analyzed using a mixed effect model with sequence, period and treatment as fixed effects and participant within sequence as a random effect; Test type: Superiority or Other; Ratio of Adjusted Means = 100.97, 90% CI 2-sided [96.28 to 105.88]

6. Secondary Outcome: Dose Normalized Area Under the Curve From Time Zero to Extrapolated Infinite Time (AUC [0-∞][dn]) for Pyrazinamide
Description: AUC [0-∞][dn] = Dose normalized area under the plasma concentration versus time curve (AUC[dn]) from time zero (pre-dose) to extrapolated infinite time (0-∞). It is obtained from AUC (0-∞) divided by dose and then multiplied by 1500. The test and reference for pyrazinamide were given at different doses, so dose-normalized parameters were used for analysis for adjusting the dose effect on bioequivalence conclusion.
Time Frame: 0 (pre-dose), 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 16, 24, 36 and 48 hrs post-dose
Population: as for outcome 2
Measure: Geometric Mean (Standard Deviation); unit: (ng*hr/mL)/mg
Arm/Group | Myrin-P Forte | Four Single Drug References
Number analyzed (Participants) | 36 | 35
(ng*hr/mL)/mg | 471000 (85153) | 464800 (92222)
Statistical Analysis 1: Comparison: Myrin-P Forte vs Four Single Drug References; Pyrazinamide; Natural log transformed AUC (0 -∞)(dn) was analyzed using mixed effect model with sequence, period and treatment as fixed effects and participant within sequence as a random effect; Test type: Superiority or Other; Ratio of Adjusted Means = 101.80, 90% CI 2-sided [99.24 to 104.43]

7. Secondary Outcome: Plasma Decay Half-life (t1/2)
Description: Plasma decay half-life is the time measured for the plasma concentration to decrease by one half.
Time Frame: 0 (pre-dose), 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 16 and 24 hrs post-dose for rifampicin, isoniazid and ethambutol and additional 36 and 48 hrs post-dose for pyrazinamide
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | Myrin-P Forte | Four Single Drug References
Number analyzed (Participants) | 36 | 35
hr
  Rifampicin (n= 36, 35) | 3.6630 (1.0477) | 3.4290 (0.6938)
  Isoniazid (n= 35, 35) | 3.7340 (0.9197) | 3.9470 (1.1751)
  Ethambutol (n= 28, 31) | 7.7430 (1.1716) | 7.6390 (1.1158)
  Pyrazinamide (n= 36, 35) | 9.8630 (1.3333) | 9.7660 (1.3671)

8. Secondary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax)
Time Frame: as for outcome 7
Population: as for outcome 2
Measure: Median (Full Range); unit: hr
Arm/Group | Myrin-P Forte | Four Single Drug References
Number analyzed (Participants) | 36 | 35
hr
  Rifampicin | 2.00 [1.00 to 4.00] | 1.50 [1.00 to 3.00]
  Isoniazid | 1.02 [0.25 to 2.52] | 1.00 [0.25 to 3.00]
  Ethambutol | 2.77 [1.00 to 4.28] | 2.48 [1.50 to 4.00]
  Pyrazinamide | 1.50 [0.25 to 3.02] | 1.50 [0.25 to 6.00]

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Myrin-P Forte | Four Single Drug References
Serious Adverse Events (participants affected / at risk) | 0/36 | 0/35
Other Adverse Events (participants affected / at risk) | 34/36 | 31/35
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Myrin-P Forte (N=36) | Four Single Drug References (N=35)
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Catheter site swelling (General disorders) | 1 | 0
Pyrexia (General disorders) | 1 | 0
Oral herpes (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Blood glucose increased (Investigations) | 1 | 1
Cardiac murmur functional (Investigations) | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 1 | 0
Chromaturia (Renal and urinary disorders) | 32 | 31
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 | 1
Drug eruption (Skin and subcutaneous tissue disorders) | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No